CLINICAL TRIAL: NCT02745483
Title: Prospective, Single-center, Single-arm, Clinical Trial Evaluating the Clinical Efficacy and Safety of a Novel Separable Cluster Electrode in Patients With Focal Liver Malignancies
Brief Title: Radiofrequency Ablation Using Octopus Electrodes for Treatment of Focal Liver Malignancies: Follow-up Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-2016-0486
Record Dates: First submitted 2016-04-05; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Separable clustered electrodes (Experimental): Enrolled patients in the prospective study (RFA using separable clustered electrodes (Octopus®)) for treatment-naive HCC (n=79)
  Interventions: Device: Separable clustered electrodes
- Historical control group (No Intervention): Patients who received RFA according to routine protocol in our center (multiple internally-cooled electrodes) for treatment-naive HCC from Jan 2011 to July 2013 in our institution (n=74) .

INTERVENTIONS:
Device: Separable clustered electrodes — patients who signed informed consent, RFA was performed using separable clustered electrodes (Octopus®) in which, inter-tine distances can be flexibly adjusted by an operator.
  Other Names: Octopus®
  Arms: Separable clustered electrodes

SUMMARY:
The purpose of this study is to compare the therapeutic outcomes and safety of the study patients who received radiofrequency ablation (RFA) using separable clustered electrodes with those of a matched historical control group who had received RFA using multiple internally-cooled electrodes.

DETAILED DESCRIPTION:
Although RFA is widely used as a curative treatment option for a variety of liver malignancies, it is generally limited for treating tumors larger than 2 cm in diameter with a sufficient tumor-free margin. Thus, various strategies are employed to create a sufficient ablation zone such as internally cooled-electrodes, expandable electrodes and adaptation of switching mono/bipolar controllers. Despite that these attempts have created larger ablative zones in clinical and preclinical studies, the efficacy should be validated in terms of clinical outcome.

In this study, investigators evaluated the therapeutic outcomes and safety of RFA using separable clustered electrodes for treatment-naive hepatocellular carcinomas (HCCs) in comparison with RFA using multiple internally-cooled electrodes. The study group is a subgroup of our prospective study cohort (NCT02683538) and a control group is a matched historical group received RFA in our institution using multiple internally-cooled electrodes.

ELIGIBILITY:
Inclusion criteria

* HCC diagnosed on biopsy OR typical imaging features of HCC on CT or MRI according to AASLD guidelines
* 1-3 HCCs equal to or smaller than 5cm in the liver
* no direct contact with or invasion into the hepatic hilar structures or inferior vena cava
* treatment-naive HCC

Exclusion criteria

* patients with uncontrolled coagulopathy
* patients with Child-Pugh classification C
* patients with tumor invasion into the portal vein or hepatic vein
* extrahepatic spread

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cumulative 1-year local tumor progression (LTP) rate | 12 months after RFA
  Comparison of rates of LTP in two groups in a year after RFA
Cumulative 2-year LTP rate | 24 months after RFA
  Comparison of rates of LTP in two groups in two years after RFA
Cumulative 3-year LTP rate | 36 months after RFA
  Comparison of rates of LTP in two groups in three years after RFA

SECONDARY OUTCOMES:
1-year Recurrence free survival rate | 12 months after RFA
  comparison of survival rate without disease progression in two groups
2-year Recurrence free survival rate | 24 months after RFA
  comparison of survival rate without disease progression in two groups
3-year Recurrence free survival rate | 36 months after RFA
  comparison of survival rate without disease progression in two groups

OTHER OUTCOMES:
Major complication rate after RFA | 30 days after RFA
  Description and comparison of the type and incidence of major complication after RFA are assessed according to Society of Interventional Radiology (SIR) grading system in two groups.
Technical success rate | 1 day after RFA
  comparison of rates of sufficient ablative zone creation which covers the whole tumor on post-RFA computed tomography (CT) in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JW, Lee JM, Lee DH, Yoon JH, Suh KS, Yoon JH, Kim YJ, Lee JH, Yu SJ, Han JK. Switching Monopolar Radiofrequency Ablation Using a Separable Cluster Electrode in Patients with Hepatocellular Carcinoma: A Prospective Study. PLoS One. 2016 Aug 30;11(8):e0161980. doi: 10.1371/journal.pone.0161980. eCollection 2016. PMID 27575787